CLINICAL TRIAL: NCT00894790
Title: A Phase IV Open Label Randomized Multicenter Comparative Study Of Celecoxib Efficacy And Safety Versus Standard Doses Of Oral Diclofenac In Acute Pain Due To Cervical Sprain Related To Motor Vehicle Accident
Brief Title: Celecoxib Efficacy And Safety Versus Diclofenac In Acute Pain Due To Cervical Sprain Related To A Traffic Accident
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A3191352
Record Dates: First submitted 2009-03-27; First posted 2009-05-07 (Estimated); Results first posted 2011-02-25 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Pain
Keywords: Treatment of the acute pain due to cervical; sprain; Celecoxib; NSAID; Diclofenac
MeSH Terms: conditions — Pain; Sprains and Strains | interventions — Celecoxib; Diclofenac

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Celecoxib
- 2 (Active Comparator)
  Interventions: Drug: oral Diclofenac

INTERVENTIONS:
Drug: Celecoxib — celecoxib 200 mg BID (twice a day) with a loading dose of 400 mg
  Arms: 1
Drug: oral Diclofenac — diclofenac 75 mg tablet BID (twice a day)
  Arms: 2

SUMMARY:
This Study Will Evaluate Celecoxib Efficacy And Safety Versus Standard Doses Of Diclofenac In Acute Pain Due To Cervical Injury (Due To A Sprain) Related To A Motor Vehicle Accident

DETAILED DESCRIPTION:
On 21Oct2010 study was prematurely terminated due to poor enrollment with subsequent low number of participants. No safety or efficacy issues were involved in the decision to terminate prematurely.

ELIGIBILITY:
Inclusion Criteria:

* Patients That Had Suffered A Car Accident And Due To It Suffered A Cervical Sprain

Exclusion Criteria:

* Recent Cervical Sprains Or Other Cervical Conditions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, México, D.F., Mexico

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191352&StudyName=Celecoxib%20Efficacy%20And%20Safety%20Versus%20%20Diclofenac%20In%20Acute%20Pain%20Due%20To%20Cervical%20Sprain%20Related%20To%20A%20Traffic%20Accident

RESULTS

PARTICIPANT FLOW:
Groups:
- Celecoxib: Celecoxib 400 mg capsules initial loading dose followed by 200 mg twice daily for up to 14 days
- Diclofenac: Diclofenac 75 mg tablets twice daily up to 14 days, according to local standard of care
Period: Overall Study
Arm/Group | Celecoxib | Diclofenac
Started | 4 | 4
Completed | 3 | 2
Not Completed | 1 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Did not meet entrance criteria | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib | Diclofenac | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Customized [Number; unit: participants]
  18 to 44 years | 2 | 2 | 4
  45 to 64 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 7 of Participant's Assessment of Cervical Pain Due to Cervical Sprain
Description: Participant rated visual analogue scale (VAS) for pain ranging from 0 to 100 mm (no pain to worst possible pain).
Time Frame: Baseline, Day 7
Population: Data not analyzed due to study termination.
Arm/Group | Celecoxib | Diclofenac
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change From Baseline on VAS-pain at Day 3 and Day 14
Description: Participant rated visual analogue scale (VAS) for pain ranging from 0 to 100 mm (no pain to worst possible pain).
Time Frame: Baseline, Days 3, 14
Population: Data not analyzed due to study termination.
Arm/Group | Celecoxib | Diclofenac
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Percentage of Participants With at Least a 20 mm Improvement on VAS-pain (Responder Rates)
Description: Participant rated visual analogue scale (VAS) for pain ranging from 0 to 100 mm (no pain to worst possible pain) with at least a 20 mm improvement.
Time Frame: Baseline, Days 7, 14
Population: Data not analyzed due to study termination.
Arm/Group | Celecoxib | Diclofenac
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change From Baseline in Patient Global Assessment of Cervical Injury
Description: Participant rated responses to question: Considering all the ways your cervical injury affects you, how are you doing today? Response options ranged from 1 (Very good - No symptoms and no limitation of normal activities) to 5 (Very Poor - Very severe symptoms which are intolerable and inability to carry out all normal activities).
Time Frame: Baseline, Days 7, 14
Population: Data not analyzed due to study termination.
Arm/Group | Celecoxib | Diclofenac
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change From Baseline on Physician's Global Assessment of Cervical Injury
Description: Physician rated responses evaluating the overall condition of participant's cervical injury at that time. Response option ranged from 1 (Very mild - Very mild signs and symptoms of cervical injury) to 5 (Very Severe - Very severe signs and symptoms of cervical injury).
Time Frame: Baseline, Days 7, 14
Population: Data not analyzed due to study termination.
Arm/Group | Celecoxib | Diclofenac
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change From Baseline in Modified Brief Pain Inventory-Short From (m-BPI-sf): Pain Interference Score
Description: m-BPI-sf: participant-rated 11 point Likert rating scale ranging from 0 (does not interfere) to 10 (completely intereres) with functional activities (general activity, mood, walking ability, relations with other people, sleep, normal work, and enjoyment of life) in past 24 hours.
Time Frame: Baseline, Days 7, 14
Population: Data not analyzed due to study termination.
Arm/Group | Celecoxib | Diclofenac
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Modified Brief Pain Inventory-Short Form (m-BPI-sf): Pain Severity Index Scores
Description: m-BPI-sf: participant rated 11-point Likert rating scale ranging from 0 (no pain) to 10 (worst pain possible). Pain severity index is the mean of item scores 2, 3, and 4 (pain right now, worst pain, and average pain level).
Time Frame: Baseline, Days 7, 14
Population: Data not analyzed due to study termination.
Arm/Group | Celecoxib | Diclofenac
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change From Baseline in Categorical Responses to Participant's Gastrointestinal (GI) Symptom Questionnaire
Description: Two part questionnaire; First part assessed symptoms: feeling of gas/air in stomach or feeling bloated, nausea, vomiting, excessive burping or belching and worsening of heartburn or acid reflux. Participant rated Yes/No experienced, for how many days per week (1 through 7) for each symptom and how bothered they were (not at all, somewhat or very). Second part assessed the presence of general abdominal pain (steady, dull, sharp/shooting, always present or comes and goes), the number of days they experienced it (1 through 7) and how bothered they were by it (not at all, somewhat, very).
Time Frame: Baseline, Days 7, 14
Population: Data not analyzed due to study termination.
Arm/Group | Celecoxib | Diclofenac
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline in Participant's Responses to Neck Disability Index (NDI)
Description: NDI: participant-administered 10-item questionnaire to assess how neck pain affects 10 activities of daily living (pain intensity, personal care, lifting, reading, headaches, concentration, work, driving, sleeping, and recreation) with six potential responses, each describing a greater degree of disability (0 = no disability to 5 = total disability). Total score calculated by adding individual item scores for evaluation scheme: 0-5 = No disability; 6-15 = Mild disability; 16-25 = Moderate disability; 26-35 = Severe disability; Above 35 = Complete disability.
Time Frame: Baseline, Days 7, 14
Population: Data not analyzed due to study termination.
Arm/Group | Celecoxib | Diclofenac
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Celecoxib | Diclofenac
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.